CLINICAL TRIAL: NCT06950541
Title: The Impact of Myofascial Therapy on Connective Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Adrian Rogala, Principal Investigator, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: JozefPilsudski_U
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Painful; Fascial Manipulation; Fascia; Pain; Myofascial Pain; Myofascial; Myofascial Dysfunction
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial therapy (Experimental)
  Interventions: Procedure: Myofascial therapy
- Deep Tissue Massage (Experimental)
  Interventions: Procedure: Deep Tissue Massage

INTERVENTIONS:
Procedure: Myofascial therapy — The myofascial therapy in the form of Fascial Distortion Model (FDM) method is based on the idea that issues within the musculoskeletal system stem from deformations or distortions in the fascia. Once the type of deformation is identified, a specific technique is employed by the physiotherapist using their hands and pressure. FDM identifies six types of fascial distortions that can cause pain and other musculoskeletal issues. These distortions include triggerbands, continuum distortions, cylinder distortions, herniated triggerpoints, tectonic fixations, and folding distortions.
  Arms: Myofascial therapy
Procedure: Deep Tissue Massage — A deep tissue massage is a therapeutic technique that focuses on realigning deeper layers of muscles and connective tissue. It is particularly beneficial for individuals dealing with chronic pain, muscle tension, or injury recovery.
  The physiotherapist uses more intense pressure compared to other massage types, like Swedish massage. The goal is to reach deeper muscle layers to relieve tension and pain. The therapist employs various techniques, including long, slow strokes, deep finger pressure, and friction, also use elbows, knuckles, or forearms to apply pressure to specific areas.
  Arms: Deep Tissue Massage

SUMMARY:
The study involved patients who suffered from myofascial pain caused occupational or sports overloads or muscle strains caused by sports or improper preparation for physical activity. The patients had not been previously treated for this reason. The only form of therapy was self-administered over-the-counter painkillers and ointments. Due to lack of relief, patients received one of two types of treatments, myofascial therapy or deep tissue massage. Each group was divided into three subgroups, depending on the location of the symptoms: arm, forearm, calf. The patients received three treatments on alternate days. Ultrasound imaging examination was performed by a physiotherapist, qualified to assess soft tissues using an USG. Two measurements were taken, before and seven days after therapy. To standardise the assessment, ultrasound imaging protocol was used.

The thickness of the fascia was measured by ImageJ software. The aim of the study was an ultrasound imaging assessment of connective tissue of patients undergone myofascial therapy.

ELIGIBILITY:
Inclusion Criteria:

* undergone myofascial therapy
* undergone deep tissue massage
* patients with pain of musculoskeletal origin
* without contraindications to myofascial therapy
* without neurological diseases
* voluntary consent to participate in the study

Exclusion Criteria:

* resignation from the study
* lack of patient consent
* cancers
* disturbed continuity of skin tissue at the examination site
* previous surgical procedures at the study site
* large vascular changes
* inflammatory changes in the examined areas of the body
* sensory disturbances in the examined body areas
* resignation from therapy
* changing the type of therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The thickness of the deep and superficial fascia. | From enrollment to the 7 days after last therapy.
  To assessed the thickness of the deep and superficial fascia, ultrasound imaging examination (USG) was performed by qualified physiotherapist. Two measurements were taken, before and seven days after therapy. Philips Affiniti 70G ultrasound device with linear probe (2-15 MHz) was used. To standardize the assessment, ultrasound imaging protocol described by Pirri et al. 2022 was used. To obtain more accurate results, the ultrasound image of the examined tissue was placed in the ImageJ ver. 1.54 software to assess the fascia thickness in millimetres.

SECONDARY OUTCOMES:
Pain level | From enrollment to the 7 days after last therapy.
  To assess the pain level, Visual Analogue Scale (VAS) was used. It is a simple but valuable instrument that measure a level of pain, by range across a continuum of values and cannot easily be directly measured. The scale is a horizontal line, 100 mm in length, anchored by word descriptors at each end, that represent the severity of symptoms from 0 "no symptoms" to 10 "very severe symptoms." The patient marked on the line the point that the patient believed represents his or her perception of his or her current state.

OTHER OUTCOMES:
Body weight | Once - upon enrollment
  A digital scale was used to assess the patients' body weight. The unit of measurement used in the study was kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pirri C, Petrelli L, Guidolin D, Porzionato A, Fede C, Macchi V, De Caro R, Stecco C. Myofascial junction: Emerging insights into the connection between deep/muscular fascia and muscle. Clin Anat. 2024 Jul;37(5):534-545. doi: 10.1002/ca.24148. Epub 2024 Mar 12. PMID 38476005
- [Background] Hughes E, Koenig J, Lee R, McDermott K, Freilicher T, Pitcher M. Pilot study assessing the effect of Fascial Manipulation on fascial densifications and associated pain. Eur J Transl Myol. 2022 Mar 3;32(1):10369. doi: 10.4081/ejtm.2022.10369. PMID 35244363
- [Background] Jha DK, Wongkaewpotong J, Chuckpaiwong B. Effect of Age and BMI on Sonographic Findings of Plantar Fascia. J Foot Ankle Surg. 2023 Jan-Feb;62(1):125-128. doi: 10.1053/j.jfas.2022.05.010. Epub 2022 May 23. PMID 35764475
- [Background] Hanson-Viana E, Rojas-Ortiz J, Rendon-Medina MA, Pacheco-Lopez RC, Rios-Lara Lopez LR, Palacios-Juarez J. Influence of BMI, Age, and Gender on the Thickness of Most Common Thinned Flaps. Plast Reconstr Surg Glob Open. 2021 Mar 30;9(3):e3409. doi: 10.1097/GOX.0000000000003409. eCollection 2021 Mar. PMID 33968546
- [Background] Kondrup F, Gaudreault N, Venne G. The deep fascia and its role in chronic pain and pathological conditions: A review. Clin Anat. 2022 Jul;35(5):649-659. doi: 10.1002/ca.23882. Epub 2022 Apr 27. PMID 35417568
- [Background] Lariviere C, Preuss R, Gagnon DH, Mecheri H, Driscoll M, Henry SM. The relationship between clinical examination measures and ultrasound measures of fascia thickness surrounding trunk muscles or lumbar multifidus fatty infiltrations: An exploratory study. J Anat. 2023 Apr;242(4):666-682. doi: 10.1111/joa.13807. Epub 2022 Dec 15. PMID 36521728
- [Background] Wilke J, Macchi V, De Caro R, Stecco C. Fascia thickness, aging and flexibility: is there an association? J Anat. 2019 Jan;234(1):43-49. doi: 10.1111/joa.12902. Epub 2018 Nov 11. PMID 30417344
- [Background] Asquini G, Pitance L, Michelotti A, Falla D. Effectiveness of manual therapy applied to craniomandibular structures in temporomandibular disorders: A systematic review. J Oral Rehabil. 2022 Apr;49(4):442-455. doi: 10.1111/joor.13299. Epub 2022 Jan 17. PMID 34931336
- [Background] Clar C, Tsertsvadze A, Court R, Hundt GL, Clarke A, Sutcliffe P. Clinical effectiveness of manual therapy for the management of musculoskeletal and non-musculoskeletal conditions: systematic review and update of UK evidence report. Chiropr Man Therap. 2014 Mar 28;22(1):12. doi: 10.1186/2045-709X-22-12. PMID 24679336
- [Background] Rogala A., Warzecha A., Turek G., Brzuszkiewicz-Kuźmicka G., Raźniak M., Dzierzęcki S., Ząbek M. The importance of manual therapy in occipital neuralgia - case study. BÓL. 2023; 24(1): 44-51. doi: 10.5604/01.3001.0053.4745.
- [Background] Rogala A., Brzuszkiewicz-Kuźmicka G. Influence of myofascial therapy on painful erection - case study. BÓL. 2020; 21(3): 54-59. doi: 10.5604/01.3001.0014.6060.
- [Background] Nunez-Cabaleiro P, Leiros-Rodriguez R. Effectiveness of manual therapy in the treatment of cervicogenic headache: A systematic review. Headache. 2022 Mar;62(3):271-283. doi: 10.1111/head.14278. Epub 2022 Mar 16. PMID 35294051
- [Background] Cumplido-Trasmonte C, Fernandez-Gonzalez P, Alguacil-Diego IM, Molina-Rueda F. Manual therapy in adults with tension-type headache: A systematic review. Neurologia (Engl Ed). 2021 Sep;36(7):537-547. doi: 10.1016/j.nrleng.2017.12.005. Epub 2020 Apr 7. PMID 34537167
- [Background] Iogna Prat P, Milan N, Huber J, Ridehalgh C. The effectiveness of nerve mechanical interface treatment for entrapment neuropathies in the limbs: A systematic review with metanalysis. Musculoskelet Sci Pract. 2024 Feb;69:102907. doi: 10.1016/j.msksp.2024.102907. Epub 2024 Jan 9. PMID 38217928
- [Background] Hyunjoong K., Seungwon L. The Impact of Manual Therapy on Pain Catastrophizing in Chronic Pain Conditions: A Systematic Review and Meta-analysis. Phys Ther Rehabil Sci. 2023; 12(2): 177-184. doi: 10.14474/ptrs.2023.12.2.177
- [Background] Tamartash H, Bahrpeyma F, Dizaji MM. The Effect of Remote Myofascial Release on Chronic Nonspecific Low Back Pain With Hamstrings Tightness. J Sport Rehabil. 2023 Mar 16;32(5):549-556. doi: 10.1123/jsr.2022-0141. Print 2023 Jul 1. PMID 36928003
- [Background] Ghorbanpour A., Shadmehr A., Moghaddam ST., Rasanani MH. The possibility of changes of brain activity following myofascial release in patients with nonspecific chronic low back pain: A hypothesis. Medical Hypotheses. 2023; 176: 111082. doi: 10.1016/j.mehy.2023.111082.
- [Background] Barassi G., Guerri S., Tavani R., Ricucci G., De Luca G., Rabini A., Di Iorio A. Ultrasonography in physiotherapy and rehabilitation. JAHC. 2021; 3(1). doi: 10.36017/jahc202131114
- [Background] Findley TW., Chaitow L., Huijing PA., Schleip R. Fascia: The Tensional Network of the Human Body. Elsevier 2012; 5 -57.
- [Background] Rogala A., Molik B., Brzuszkiewicz-Kuźmicka G., Truszczyńska-Baszak A. The impact of Fascial Distortion Model on Shoulder Girdle Dysfunction. Med Rehabil 2022; 26(2): 17-26. doi: 10.5604/01.3001.0015.8242
- [Background] Baird CJ., Shumate SM., Tancredi MP., Cayce LM., Wibbenmeyer JL. The effects of the fascial distortion model on chronic hamstring tightness. Topics in Integrative Health Care. 2014; 6(2): 1074-1086.
- [Background] LeeChan JK., Kim M. Comparison of Maximum Isometric Strength, Proprioceptive, Dynamic Balance, and Maximum Angle by Applying the Fascial Distortion Model to Chronic Ankle Instability Subjects. J Kor Phys Ther. 2021; 33(5): 224-230. doi: 10.18857/jkpt.2021.33.5.224
- [Background] Ghorbanpour A. Fascial Treatment in Frozen Shoulder: A Case Report. Journal of Modern Rehabilitation. 2019; 13(2): 123-128. doi: 10.32598/JMR.13.2.123
- [Background] Tozzi P., Chila A., Liem T. Fascia in the Osteopathic Field. Handspring Publishing Limited. 2017; 35: 360 -367
- [Background] Schulze C, Finze S, Bader R, Lison A. Treatment of medial tibial stress syndrome according to the fascial distortion model: a prospective case control study. ScientificWorldJournal. 2014;2014:790626. doi: 10.1155/2014/790626. Epub 2014 Oct 14. PMID 25379543
- [Background] Stecco C, Pirri C, Fede C, Fan C, Giordani F, Stecco L, Foti C, De Caro R. Dermatome and fasciatome. Clin Anat. 2019 Oct;32(7):896-902. doi: 10.1002/ca.23408. Epub 2019 May 28. PMID 31087420
- [Background] Pirri C, Stecco C, Petrelli L, De Caro R, Ozcakar L. Reappraisal on the Superficial Fascia in the Subcutaneous Tissue: Ultrasound and Histological Images Speaking Louder Than Words. Plast Reconstr Surg. 2022 Jul 1;150(1):244e-245e. doi: 10.1097/PRS.0000000000009224. Epub 2022 May 24. No abstract available. PMID 35608834
- [Background] Pirri C, Stecco C, Pirri N, De Caro R, Ozcakar L. Ultrasound examination for a heel scar: seeing/treating the painful superficial fascia. Med Ultrason. 2022 May 25;24(2):255-256. doi: 10.11152/mu-3689. PMID 35617618
- [Background] Pirri C, Pirri N, Guidolin D, Macchi V, De Caro R, Stecco C. Ultrasound Imaging of the Superficial Fascia in the Upper Limb: Arm and Forearm. Diagnostics (Basel). 2022 Aug 4;12(8):1884. doi: 10.3390/diagnostics12081884. PMID 36010234
- [Background] Pirri C, Guidolin D, Fede C, Macchi V, De Caro R, Stecco C. Ultrasound Imaging of Brachial and Antebrachial Fasciae. Diagnostics (Basel). 2021 Dec 2;11(12):2261. doi: 10.3390/diagnostics11122261. PMID 34943498
- [Background] Pirri C, Stecco A, Fede C, De Caro R, Stecco C, Ozcakar L. Ultrasound imaging of a scar on the knee: Sonopalpation for fascia and subcutaneous tissues. Eur J Transl Myol. 2020 Apr 1;30(1):8909. doi: 10.4081/ejtm.2019.8909. eCollection 2020 Apr 7. PMID 32499900
- [Background] Pirri C, Stecco C, Fede C, Macchi V, Ozcakar L. Ultrasound Imaging of the Fascial Layers: You See (Only) What You Know. J Ultrasound Med. 2020 Apr;39(4):827-828. doi: 10.1002/jum.15148. Epub 2019 Oct 23. No abstract available. PMID 31642543
- [Background] Pirri C, Fede C, Stecco A, Guidolin D, Fan C, De Caro R, Stecco C. Ultrasound Imaging of Crural Fascia and Epimysial Fascia Thicknesses in Basketball Players with Previous Ankle Sprains Versus Healthy Subjects. Diagnostics (Basel). 2021 Jan 26;11(2):177. doi: 10.3390/diagnostics11020177. PMID 33530583
- [Background] Boucher JD, Figueroa J. Restoration of Full Shoulder Range of Motion After Application of the Fascial Distortion Model. J Am Osteopath Assoc. 2018 May 1;118(5):341-344. doi: 10.7556/jaoa.2018.044. PMID 29507951
- [Background] Richter D, Karst M, Buhck H, Fink MG. Efficacy of Fascial Distortion Model Treatment for Acute, Nonspecific Low-Back Pain in Primary Care: A Prospective Controlled Trial. Altern Ther Health Med. 2017 Sep;23(5):AT5522. Epub 2017 Jun 23. PMID 28646809
- [Background] Chaudhry H, Schleip R, Ji Z, Bukiet B, Maney M, Findley T. Three-dimensional mathematical model for deformation of human fasciae in manual therapy. J Am Osteopath Assoc. 2008 Aug;108(8):379-90. doi: 10.7556/jaoa.2008.108.8.379. PMID 18723456
- [Background] Thalhamer C. A fundamental critique of the fascial distortion model and its application in clinical practice. J Bodyw Mov Ther. 2018 Jan;22(1):112-117. doi: 10.1016/j.jbmt.2017.07.009. Epub 2017 Jul 25. PMID 29332733
- See also: Anatomy, Fascia Layers; 2023 — https://www.ncbi.nlm.nih.gov/books/NBK526038/